CLINICAL TRIAL: NCT00538278
Title: Prospective Database for Acute Myeloblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RAC #2051-057
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Leukemia, Myeloblastic, Acute
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Database Management Systems; Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — database
  Other Names: Registry

SUMMARY:
Prospective Database for Acute Myeloblastic Leukemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Chaudhri, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center